CLINICAL TRIAL: NCT05004662
Title: Partnering With a State Food Bank to Provide Tobacco Treatment to Underserved Smokers (Project NOURISH)
Brief Title: Partnering With Food Bank to Provide Tobacco Treatment to Underserved Smokers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MCC-20154; 5R01CA231952-03 (NIH)
Record Dates: First submitted 2021-08-06; First posted 2021-08-13 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Treatment (Active Comparator): Participants randomized to Standard Treatment (ST) will be provided with a 10-week supply of nicotine patches and lozenges. ST participants will be connected with Florida Quitline services and will complete weekly 4-item smartphone assessments electronically for 26 weeks. The weekly assessments consist of questions on smoking status, motivation, self-efficacy, and perceived stress.
  Interventions: Drug: Nicotine patch; Behavioral: Counceling; Drug: Nicotine lozenge
- Automated Treatment (Experimental): Participants randomized to Automated Treatment (AT) will be given a 10-week supply of nicotine patches and lozenges. AT will also comprise of: 1) 12 proactive treatment videos, delivered weekly, that are tailored on smoking status, motivation, agency, and/or negative affect/stress; 2) 26 weeks of on-demand access to treatment content; 3) 26 weeks of text content
  Interventions: Behavioral: Smartphone-delivered automated treatment; Drug: Nicotine patch; Drug: Nicotine lozenge

INTERVENTIONS:
Behavioral: Smartphone-delivered automated treatment — An interactive smartphone-based intervention that comprises content delivered via audio/video clips and text content automatically each week to the participant
  Arms: Automated Treatment
Drug: Nicotine patch — Participants will be provided with a 10-week supply of nicotine patches
Behavioral: Counceling — Phone counseling with the Florida Quitline
  Arms: Standard Treatment
Drug: Nicotine lozenge — Participants will be provided with a 10-week supply of nicotine lozenges

SUMMARY:
This study will evaluate the efficacy and economic impact of a theoretically-based, fully automated, interactive smartphone-based smoking cessation intervention.

ELIGIBILITY:
Inclusion Criteria:

* >100 lifetime cigarettes
* English or Spanish speaking
* Currently smoke > 5 cigarettes/day
* Process a smartphone compatible with the project app
* Have a valid email address

Exclusion Criteria:

* Currently pregnant or breastfeeding
* Current use of smoking cessation medications
* Enrolled in a smoking cessation study
* Household member enrolled in the study
* Failure to electronically confirm participation with 14 days of randomization via electronic link sent to participant's smartphone

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 520 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2026-06-03 (Estimated)

PRIMARY OUTCOMES:
Self Reported 7 Day Abstinence Smoking Status | 12 Month Follow-Up
  Participants will self report 7-day abstinence smoking status

SECONDARY OUTCOMES:
Smoking Status by Saliva Cotinine Kit | 12 Month Follow-Up
  Investigators will verify smoking status by collecting cotinine sample from a saliva cotinine kit.
Self Reported 24 Hours Smoking Abstinence | 12 Month Follow-Up
  Number of participants who report they quit smoking for 24 hours
30 Day Smoking Abstinence | 12 Month Follow-Up
  Number of participants who report they quit smoking for 30 days
Continuous Smoking Abstinence | 12 Month Follow-Up
  Number of participants who report they quit smoking

CONTACTS AND LOCATIONS:
Overall Officials: Damon J Vidrine, Dr.PH, Principal Investigator — Moffitt Cancer Center; Jennifer I Vidrine, Ph.D., Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vidrine JI, Shih YT, Businelle MS, Sutton SK, Hoover DS, Cottrell-Daniels C, Fennell BS, Bowles KE, Vidrine DJ. Comparison of an automated smartphone-based smoking cessation intervention versus standard quitline-delivered treatment among underserved smokers: protocol for a randomized controlled trial. BMC Public Health. 2022 Mar 22;22(1):563. doi: 10.1186/s12889-022-12840-7. PMID 35317789
- See also: Moffitt Cancer Center Clinical Trial Search — https://www.moffitt.org/clinical-trials-research/clinical-trials/?gclid=EAIaIQobChMImIymzIa-9gIVAZ2GCh3uzAWJEAAYASAAEgI0ovD_BwE